CLINICAL TRIAL: NCT05790616
Title: Accuracy of Pulse Oximeters During Profound Hypoxia
Acronym: APO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ITS_002
Record Dates: First submitted 2023-02-10; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hypoxia
Keywords: SpO2; photoplethysmography; camera based photoplethysmography
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NI(Fast-Sitting) (Experimental): Subgroup Non-Invasive (Fast-Sitting): sitting volunteers undergo an ambient oxygen decrease from 21% to 10% (SpO2 <73% for 1 minute) followed by a fast increase of ambient oxygen concentration.
  Fast: if the study is completed for a volunteer reaching SpO2 ≤73%, the subject leaves the room and breaths 21% oxygen. The hypoxia inducing device is stopped after all subjects left the hypoxia room and the door of the hypoxia room is opened, allowing air with 21% O2 to enter the room. Airco fan stays running.
  Interventions: Other: Oxygen reduction
- NI(Slow-Sitting) (Experimental): Volunteers of subgroup Non-Invasive (Slow-Sitting) follow the NI (Rapid-Sitting) protocol, but after hypoxia at FiO2=0,10 oxygen normalization is programmed to increase at the same speed as the hypoxia creation.
  Slow: after target hypoxia has been reached, air with 21% of oxygen is allowed to enter the room in such a way that the speed of increase of O2 to 21% is approximately equal to the decrease of the room's oxygen to 10%
  Interventions: Other: Oxygen reduction
- NI(Fast-Lying) (Experimental): Volunteers included in the Non-Invasive (Fast-Lying) group follow the NI (Rapid-sitting) protocol although in lying position.
  Interventions: Other: Oxygen reduction
- IN(Fast-Sitting) (Experimental): After full completion of the Non-Invasive (NI) studies, and a defined algorithm to compute SpO2 by TDw1 is achieved, the study is repeated as described for the NI (Rapid-Sitting) protocol, but arterial blood oxygen saturation (SaO2) will be determined during 5 stable ambient oxygen plateaus (the Invasive (Fast-Sitting) study). These results are used as benchmark to define the final accuracy of TDw1 for SpO2 reproduction. In this part of the study, according to the minimal requirements of the regulatory agencies, 12 volunteers that successfully completed the study will be included.
  Interventions: Procedure: Arterial blood draw; Other: Oxygen reduction

INTERVENTIONS:
Procedure: Arterial blood draw — For the IN(Fast-Sitting) arm arterial blood will be collected to derive "Gold-standard" SaO2 reference values.
  Arms: IN(Fast-Sitting)
Other: Oxygen reduction — Volunteers undergo an ambient oxygen decrease from 21% to 10%

SUMMARY:
This study is designed to calibrate and determine the accuracy for SpO2, pulse rate and respiratory rate of the newly in-house build Test Device wrist 1 (TDw1, or EVA) at Philips.

SpO2, pulse rate and respiratory rate during hypoxia will be calculated by using data of well-known reference devices, including:

* A reference SpO2 sensor of Nellcor placed at a fingertip, that reflects also continuously the pulse rate Will be used to compare with the test device.
* A reference respiratory rate device that calculates the respiratory rate based on detection of end-tidal CO2 peaks by capnography.
* Oxygen saturation in arterial blood samples (SaO2), determined by a co-oximeter will be used to calculate the accuracy of the test device.

During the study the following devices will be additionally used by the volunteers:

* AppleWatch 7
* TDw2, watch build by philips, using the PPG and software technology developed by Philips
* A smartphone that detects reflected PPG signals from the reflected screen at the handpalm, by the build in frontfacing camera (TDc) of the smartphone

Volunteers will undergo progressive hypoxia (9 min/% O2) from 21 to 10% O2 in an altitude room, resulting in a volunteer's SpO2 of 73%. During this deliberated hypoxia, the volunteers wear the test and reference devices.

This study consists of 4 sub-studies (NI = non-invasive; IN = invasive with an arterial line):

* NI (Fast-Sitting): volunteers are seated in the hypoxia room in which the ambient oxygen concentration decreases at a speed of 9 min/% O2. If the volunteer reached a SpO2 ≤73% for more than 1 minute, he/she leaves the hypoxia room. And will breath air with 21% oxygen. Volunteers wear TDw1 and TDw2 and the reference devices.
* NI(Fast-Lying): identical to NI(Fast-Sitting) but volunteers lay on a mattress. Volunteers wear TDw1 and AppleWatch 7 and the reference devices.
* NI (Slow-Sitting): identical to NI (Fast-Sitting), but after one of the volunteers reaches a SpO2 ≤73% for more than one minute, oxygen in the room increases at a speed of 9 min/% O2 until normal ambient air oxygen concentration of 21%. Volunteers wear TDw1 and AppleWatch 7 and the reference devices.
* IN(Fast-Sitting): identical to NI(Fast-Sitting) but the volunteer's oxygen saturation in blood samples withdrawn via an arterial line is measured in the laboratory.

The NI studies include 18 healthy participants in each sub-study. After the first volunteers have completed the study, small adaptations in the software of the study devices is still possible, e.g. to increase the quality of the PPG-signals. After the three sub-studies are completed, the algorithm for conversion of raw PPG signals to SpO2, pulse rate and respiratory rate will be defined and fixed for the test devices.

During the IN-study, which can only be started after completion of all NI studies, an arterial catheter will be inserted in the radial artery of the 12 participating volunteers, in order to take several blood samples to measure oxygen saturation in the blood (25 samples at well-defined moments during the study per volunteer). Using these results of arterial oxygen saturation, the accuracy of the test devices can be calculated.

ELIGIBILITY:
Inclusion Criteria:

• Healthy subjects (ASA 1 and ASA 2) between 18 and 65 years of age upon signing the informed consent. (ASA: American Society of Anesthesiologist's health score). In each group, at least 30% of one gender need to be present, and at least 15% of participants have a Fitzpatrick's skin color scale of 5 or 6.

Exclusion Criteria:

* Heavy smokers or individuals exposed to high levels of carbon monoxide that result in elevated carboxyhemoglobin levels.
* Individuals subject to conditions that result in elevated levels of methemoglobin.
* Individuals with low SpO2 or SaO2 (<95%) at FiO2 = 0,21
* Moderate to severe claustrophobia for small rooms
* Severe obesity (BMI > 35 kg/m2)
* Hemoglobinopathies
* Arteriopathies, including Raynaud disease
* ASA 3 to 5 subjects
* Tattoo's, skin lesions,use of skin lotions or use of nail polish/fake nails at the region of interest for TDw and TDc
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Algorithm validation | 90 minutes per test per participant
  1. the calculation and validation of the algorithm for
     1. conversion of the modulation ratio R of theraw PPG signals to SpO2 for all wrist Test Devices.
     2. conversion of PPG signals to PR and RR.
  2. determining the accuracy of TDw1 and TDc with cooximetry as golden benchmark in the IN study.
  3. Looking for the feasibility of TDw2 for further development
  The accuracy is represented by A(rms), and specifically for the NI study, the SpO2 range is continuous (SpO2 100- 73%, about 16 000 samples per volunteer). During the IN study the accuracy is represented by A(rms) and calculated for SpO2 versus Sa O2 (about 20 to 25 samples per volunteer).

SECONDARY OUTCOMES:
Plateau 1 | 90 minutes per test per participant
  Bias and 95% limits of agreement (LOA) of TDw1 SpO2 - Nellcor SpO2 in 90-100% Nellcor SpO2 range
Plateau 2 | 90 minutes per test per participant
  Bias and 95% LOA of TDw1 SpO2 - Nellcor SpO2 in 80-90% Nellcor SpO2 range
Plateau 3 | 90 minutes per test per participant
  Bias and 95% LOA of TDw1 SpO2 - Nellcor SpO2 in 70-80% Nellcor SpO2 range
Plateau 4 | 90 minutes per test per participant
  Bias and 95% LOA of TDw1 SpO2 - Nellcor SpO2 in 70-100% Nellcor SpO2 range
Statistics pooled subjects | 90 minutes per test per participant
  Bland-Altman of pooled subjects' TDw1 SpO2 - Nellcor SpO2
Statistics individual subject | 90 minutes per test per participant
  Bland-Altman of Bias for each individual subject
Statistics individual subject 2 | 90 minutes per test per participant
  Line listing for each individual subject

CONTACTS AND LOCATIONS:
Overall Officials: Raf De Jongh, MD, Principal Investigator — Hypoxia Centre of the Complementary Medical Centre (CMC) Genk
Locations (1):
- Hypoxia Centre of the Complementary Medical Centre (CMC), Genk, Belgium

IPD SHARING:
Plan to Share IPD: No